CLINICAL TRIAL: NCT02012309
Title: Mechanisms of Impaired HIV-associated B Cell and Pneumococcal Vaccine Responses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-2405; R01AI108479 (NIH)
Record Dates: First submitted 2013-12-10; First posted 2013-12-16 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: HIV; Pneumococcal Infections; Pneumococcal Vaccines
Keywords: HIV; Streptococcus pneumoniae infection; Streptococcus pneumoniae colonization; Pneumococcal vaccines; Prevnar; Pneumovax; Nasopharyngeal microbiome
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine; Heptavalent Pneumococcal Conjugate Vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HIV-seronegative (Experimental): HIV-seronegative subjects will receive Prevnar (PCV-13) at week 0.
  Interventions: Biological: PCV-13
- HIV-infected (Experimental): HIV-infected subjects will receive Prevnar (PCV-13) at week 0, and Pneumovax (PPSV-23) at week 8 per Advisory Committee on Immunization Practices (ACIP) guidelines.
  Interventions: Biological: PCV-13; Biological: PPSV-23

INTERVENTIONS:
Biological: PCV-13
  Other Names: Prevnar
Biological: PPSV-23
  Other Names: Pneumovax
  Arms: HIV-infected

SUMMARY:
Human Immunodeficiency Virus (HIV) infection is complicated by high rates of infections and cancers which are often the cause of death rather than the HIV/acquired immune deficiency syndrome (AIDS) virus itself. Treatment of HIV with antiretroviral medications has decreased the frequency of many complications by over 90%, but bacterial pneumonia remains extremely high. Current vaccines are not very effective in preventing these infections in patients with HIV infection. The investigators are studying the cells (B cells) that make antibodies to fight infection by binding to and killing bacteria. The goal is to understand how HIV impairs the ability of B cells to make antibodies in sufficient quantity and of sufficient quality to protect patients with HIV to learn how to enhance protection against these infections. The investigators also seek to understand the role of the bacteria (specifically Streptococcus pneumoniae) that normally live in the nose and throat in the development of pneumonia and other infections.

ELIGIBILITY:
Inclusion Criteria:

For HIV-infected subjects:

* adults aged 18-55 years
* >200 CD4+ T-cells/microliter
* no antiretroviral therapy (at the time of nasal swab/week 0)
* receiving antiretroviral therapy for >6 weeks (at the time of vaccination/week 12)

For HIV-seronegative controls:

* adults aged 18-55 years

Exclusion Criteria:

For all subjects:

* age <18 or >55 years
* history of prior pneumococcal vaccination
* immunosuppressive therapy, defined as: prednisone >15mg/day currently or >14 days in the past 3 months, cytotoxic agents, anti-metabolites, cyclosporine, anti-tumor necrosis factor, B cell monoclonal antibodies
* current or chronic pulmonary infection (bacterial, fungal, mycobacterial), pneumonia, or rhinosinusitis within 2 months
* chronic lung disease
* renal insufficiency, defined as serum creatinine >1.6
* active liver disease, including hepatitis C virus infection
* history of splenectomy
* history of antibacterial therapy within 3 months of nasal swab (week 0)
* current alcohol abuse
* chronic heart disease
* diabetes
* current cigarette smoking

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
B and T cell subsets | Weeks -12, 0, 1, 8, 9, 16
  Activation and subset distribution of B and T cell subsets and cluster of differentiation positive (CD4+) T cells and T follicular helper (TFH) cells on days 0 and 7 after stimulation
Total IgG, IgM and IgA | Weeks -12, 0, 1, 8, 9, 16
  Total immunoglobulin G (IgG), immunoglobulin M (IgM) and immunoglobulin A (IgA) produced from culture of peripheral blood mononuclear cells (PBMC) stimulated in triplicate with B cell stimuli on day 7 by enzyme-linked immunosorbent assay (ELISA)
Antibody-secreting cells | Weeks 0, 1, 8, 9
  Total IgG, IgM and IgA antibody-secreting cells (ASC) enumerated by enzyme-linked immunospot (ELISPOT) on day 0 and day 7
AID and BCL-6 production | Weeks -12, 0, 1, 8, 9, 16
  RNA extraction for activation-induced cytidine deaminase (AID) and B cell lymphoma protein 6 (BCL6) expression and mutation from stimulated B cells

SECONDARY OUTCOMES:
S.pneumoniae colonization and nasopharyngeal microbiome | Weeks -12, 0, 8, 16
  Prevalence of nasopharyngeal S. pneumoniae determined by quantitative polymerase chain reaction(Q-PCR) and 16S ribosomal RNA (rRNA) sequencing, related microbiota (commensal bacteria) and correlation between colonization and levels of pneumococcal capsule-specific IgG
S.pneumoniae urine antigen positivity | Week -12
  S. pneumoniae urine antigen positivity in relation to colonization

CONTACTS AND LOCATIONS:
Overall Officials: Edward N Janoff, MD, Principal Investigator — University of Colorado-Denver, Denver VA Medical Center
Locations (3):
- United States (3):
  - University of Colorado-Denver, Aurora, Colorado
  - Denver Health and Hospitals, Denver, Colorado
  - Denver VA Medical Center, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No